CLINICAL TRIAL: NCT03783637
Title: Measuring Single-Serving Grain Intake
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: USDA Beltsville Human Nutrition Research Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Janet Novotny, Research Physiologist, USDA Beltsville Human Nutrition Research Center
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: HS62 - Single Grain
Record Dates: First submitted 2018-12-11; First posted 2018-12-21 (Actual); Last update posted 2019-07-05 (Actual); Status verified 2019-07

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Whole Grain Oat (Other): Volunteers will consume a breakfast meal containing whole grain oats after 7 days of a whole grain free diet.
  Interventions: Other: Whole grain oats
- Whole Grain Wheat (Other): Volunteers will consume a breakfast meal containing whole grain wheat after 7 days of a whole grain free diet.
  Interventions: Other: Whole grain wheat

INTERVENTIONS:
Other: Whole grain oats — A meal containing whole grain oats
  Arms: Whole Grain Oat
Other: Whole grain wheat — A meal containing whole grain wheat
  Arms: Whole Grain Wheat

SUMMARY:
The primary objective of this study is to identify markers of a single meal of whole grain oat and whole grain wheat intake in humans.

DETAILED DESCRIPTION:
The aim of this study is to identify compounds that are found in blood and urine and are derived from a single meal of whole grain oat or whole grain wheat intake so that epidemiological studies can be conducted to provide more accurate associations between whole grain intake and health.

ELIGIBILITY:
Inclusion Criteria:

* 21 to 75 years of age
* Voluntarily agree to participate and sign an informed consent form

Exclusion Criteria:

* Body weight less than 110 lbs.
* Have a body mass index below 19 or above 38 kg/m2
* Known (self-reported) allergy or adverse reaction to study foods
* Women who have given birth during the previous 12 months or who are pregnant/lactating or who plan to become pregnant during the study
* History of bariatric surgery or nutrient malabsorption disease (such as celiac disease), Crohn's disease, diabetes, or metabolic disorders that may interfere with the study
* History of certain cancer diagnosis or treatment in the last 3 years
* Smoking or use of tobacco products in the past 6 months
* Suspected or known strictures, fistulas or physiological/mechanical GI obstruction
* Use of certain medications or supplements (prescription or over-the-counter) that may interfere with the study objectives, including blood thinning medications
* Unable or unwilling to give informed consent or communicate with study staff
* Self-report of alcohol or substance abuse within the past 12 months and/or current treatment for these problems (long-term participation in Alcoholics Anonymous is not an exclusion)
* Other medical, psychiatric, or behavioral factors that in the judgment of the Principal Investigator may interfere with study participation or the ability to follow the intervention protocol

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2019-05-13 (Actual); Primary Completion 2019-06-19 (Actual); Study Completion 2019-06-19 (Actual)

PRIMARY OUTCOMES:
Identification of unknown biomarkers of grain intake immediately after grain consumption | Day 8
  Blood and Urine metabolomics profiling will be conducted. Metabolomics refers to the complete set of small molecule metabolites. The METLIN Metabolomics Database is a repository of such chemicals and contains over 75,000 entries, thus metabolomics is a very broad assessment. Blood and urine will be broadly analyzed with mass spectrometers for metabolomics, and all ionizing compounds will be captured by the detector, which reports the ratio of mass of the compound to the charge (units: m/z which is mass to charge). The mass-to-charges will be compared across different time points of collection, and appearance of mass-to-charges in some collections (but not found in others when grains were not consumed) will indicate a biomarker of grain intake.
Identification of unknown biomarkers of grain intake a day after grain consumption | Day 9
  Blood and Urine metabolomics profiling will be conducted. Metabolomics refers to the complete set of small molecule metabolites. The METLIN Metabolomics Database is a repository of such chemicals and contains over 75,000 entries, thus metabolomics is a very broad assessment. Blood and urine will be broadly analyzed with mass spectrometers for metabolomics, and all ionizing compounds will be captured by the detector, which reports the ratio of mass of the compound to the charge (units: m/z which is mass to charge). The mass-to-charges will be compared across different time points of collection, and appearance of mass-to-charges in some collections (but not found in others when grains were not consumed) will indicate a biomarker of grain intake.
Identification of unknown biomarkers of grain intake 2 days after grain consumption | Day 10
  Urine metabolomics profiling will be conducted. Metabolomics refers to the complete set of small molecule metabolites. The METLIN Metabolomics Database is a repository of such chemicals and contains over 75,000 entries, thus metabolomics is a very broad assessment. Urine will be broadly analyzed with mass spectrometers for metabolomics, and all ionizing compounds will be captured by the detector, which reports the ratio of mass of the compound to the charge (units: m/z which is mass to charge). The mass-to-charges will be compared across different time points of collection, and appearance of mass-to-charges in some collections (but not found in others when grains were not consumed) will indicate a biomarker of grain intake.
Identification of unknown biomarkers of grain intake immediately after grain consumption | Day 34
  Blood and Urine metabolomics profiling will be conducted. Metabolomics refers to the complete set of small molecule metabolites. The METLIN Metabolomics Database is a repository of such chemicals and contains over 75,000 entries, thus metabolomics is a very broad assessment. Blood and urine will be broadly analyzed with mass spectrometers for metabolomics, and all ionizing compounds will be captured by the detector, which reports the ratio of mass of the compound to the charge (units: m/z which is mass to charge). The mass-to-charges will be compared across different time points of collection, and appearance of mass-to-charges in some collections (but not found in others when grains were not consumed) will indicate a biomarker of grain intake.
Identification of unknown biomarkers of grain intake a day after grain consumption | Day 35
  Blood and Urine metabolomics profiling will be conducted. Metabolomics refers to the complete set of small molecule metabolites. The METLIN Metabolomics Database is a repository of such chemicals and contains over 75,000 entries, thus metabolomics is a very broad assessment. Blood and urine will be broadly analyzed with mass spectrometers for metabolomics, and all ionizing compounds will be captured by the detector, which reports the ratio of mass of the compound to the charge (units: m/z which is mass to charge). The mass-to-charges will be compared across different time points of collection, and appearance of mass-to-charges in some collections (but not found in others when grains were not consumed) will indicate a biomarker of grain intake.
Identification of unknown biomarkers of grain intake 2 days after grain consumption | Day 36
  Urine metabolomics profiling will be conducted. Metabolomics refers to the complete set of small molecule metabolites. The METLIN Metabolomics Database is a repository of such chemicals and contains over 75,000 entries, thus metabolomics is a very broad assessment. Urine will be broadly analyzed with mass spectrometers for metabolomics, and all ionizing compounds will be captured by the detector, which reports the ratio of mass of the compound to the charge (units: m/z which is mass to charge). The mass-to-charges will be compared across different time points of collection, and appearance of mass-to-charges in some collections (but not found in others when grains were not consumed) will indicate a biomarker of grain intake.

SECONDARY OUTCOMES:
Blood glucose | Days 8 and 34
  Blood glucose will be measured. Blood glucose is reported in mmol/L.
Serum insulin | Days 8 and 34
  Serum insulin will be measured. Serum insulin is reported in mIU/L.
Serum c-peptide | Days 8 and 34
  Serum c-peptide will be measured. Serum c-peptide is reported in ng/ml.
Non-esterified fatty acids in blood | Days 8 and 34
  Non-esterified fatty acids will be measured in blood. Non-esterified fatty acids are reported as mEQ/L.
Triglycerides in blood | Days 8 and 34
  Triglycerides will be measured. Triglycerides are reported as mmol/L.

CONTACTS AND LOCATIONS:
Locations (1):
- USDA-ARS Beltsville Human Nutrition Research Center, Beltsville, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Li Y, Novotny JA, Baer D, Hu Y, Sun Q, Zhang S, Sang S. Betainized metabolites as biomarkers of whole grain wheat, not oat: insights from controlled crossover pharmacokinetic and daily feeding studies. Am J Clin Nutr. 2025 Dec 19:101139. doi: 10.1016/j.ajcnut.2025.101139. Online ahead of print. PMID 41423132